CLINICAL TRIAL: NCT01720082
Title: Randomized Controlled Trial Comparing Single Incision Laparoscopic Appendectomy Versus Standard Three Port Appendectomy in a Selected Cohort of Patients
Brief Title: Laparoscopic Appendectomy by Multi-port vs Single Port.
Acronym: AMUSING
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Associazione Chirurghi Ospedalieri Italiani (Other)
Collaborators: Società Italiana di Chirurgia Endoscopica e nuove tecnologie (SICE) (Unknown)
Responsible Party: Principal Investigator, Nereo Vettoretto, MD, Associazione Chirurghi Ospedalieri Italiani
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACOI - SICE
Record Dates: First submitted 2012-10-31; First posted 2012-11-02 (Estimated); Last update posted 2012-11-05 (Estimated); Status verified 2012-11

CONDITIONS: Acute Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single incision laparoscopic appendectomy (Active Comparator): Acute appendicitis with surgical indication
  Interventions: Procedure: Single incision laparoscopic appendectomy
- Multiport Laparoscopic appendectomy (Active Comparator): Acute appendicitis with surgical indication
  Interventions: Procedure: Multiport laparoscopic appendectomy

INTERVENTIONS:
Procedure: Single incision laparoscopic appendectomy — A multiport device will be introducted through a 2-2.5 transumbilical incision. Retraction of the appendix would be performed with a forceps. The mesoappendix will be divided with bipolar or monopolar cautery. The appendix stump will be ligated with suture loop or with an endo-stapler. The specimen will be delivered within a plastic bag or in any protected way (without any contact with the abdominal wall) via the umbilical port. Any fluid will be suctioned and washing performed if required. Fascial defects will be closed with 2-O polydioxanone sutures and skin closed with 4-O non-absorbable sutures. No pelvic drain will be inserted. A three-band dressing will be applied in the end.
  Other Names: SILA
  Arms: Single incision laparoscopic appendectomy
Procedure: Multiport laparoscopic appendectomy — Three ports will be inserted as follows: One 10/12 umbilical port, one 5mm suprapubic (or right suprapubic)port, one 5mm or 10/12mm port in left iliac fossa (or left suprapubic). One additional trocar can be inserted following surgeons preference. Retraction of the appendix would be performed with a forceps. The mesoappendix will be divided with bipolar or monopolar cautery. The appendix stump will be ligated with suture loop or with an endo-stapler. The specimen will be delivered within a plastic bag or in any protected way (without any contact with the abdominal wall) via the umbilical port. Any fluid will be suctioned and washing performed if required. Fascial defects (10/12 trocars)will be closed with 2-O polydioxanone sutures and skin closed with 4-O non-absorbable sutures. No pelvic drain will be inserted. A three-band dressing will be applied in the end.
  Other Names: LA
  Arms: Multiport Laparoscopic appendectomy

SUMMARY:
Laparoscopic appendectomy (LA) is nowadays considered the gold standard in fertile women affected by uncomplicated appendicitis. The level of evidence for benefits from LA in this subgroup is high. Since the dissemination of single access surgery (no-scars surgery) ameliorated outcome has been supposed in these patients regarding post-operative pain, hospital stay and cosmetics results, and keeping the same safety as LA. This randomized controlled study is supposed to give answers to these questions.

ELIGIBILITY:
Inclusion Criteria:

* age: 14-60
* American Society of Anesthesiologists (ASA) score: I-III
* absence of non-correctable coagulopathy (international normalized ratio >1,5, or platelet count <90 × 109/l).
* diagnosis: acute appendicitis with surgical indication

Exclusion Criteria:

* Complicated appendicitis after exploration or previously diagnosed (CT)
* Psychical inability
* Pregnancy

Ages: 14 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-08 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Morbidity and mortality | 30 days

SECONDARY OUTCOMES:
Post-operative pain score | 3 days
  Visual Analogic Scale (VAS scale)
Operative time | 1 day
Cosmetic result | 6 months
  VAS scale
Post-operative hospital stay | 7 days
Incision related morbidity | 6 months
  during hospital stay (7days): infectious morbidity during follow-up (6 months): incisional hernias
Quality of life | 6 months
  Gastro Intestinal Quality of Life Index (GIQLI) score at discharge and at 6 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nereo Vettoretto, MD, Study Chair — ACOI - SICE; Ferdinando Agresta, MD, Study Chair — ACOI - SICE; Luigi Boni, MD, FACS, Study Chair — SICE
Locations (1):
- M.Mellini Hospital, Chiari, BS, Italy